CLINICAL TRIAL: NCT01531569
Title: Community Alliance for Quality of Life in Long Term Care: Single Oral Dose of BeneFlax to Healthy Young and Older Adults
Brief Title: Single Oral Dose of BeneFlax to Healthy Young and Older Adults
Acronym: SOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Jane Alcorn, Ph.D., University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NHPD - 174041
Record Dates: First submitted 2012-01-09; First posted 2012-02-13 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2; Hypercholesterolemia
Keywords: Flaxseed; Lignans; Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia | interventions — secoisolariciresinol diglucoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BeneFlax (Experimental): BeneFlax given as a single oral dose to assess pharmacokinetics
  Interventions: Other: BeneFlax - 38% secoisolariciresinol diglucoside (SDG)

INTERVENTIONS:
Other: BeneFlax - 38% secoisolariciresinol diglucoside (SDG) — 0.8g of BeneFlax (contains 300mg SDG) given once by mouth
  Other Names: Secoisolariciresinol diglucoside (SDG)

SUMMARY:
This study is being done to look at age differences in the way the investigators bodies break down a compound found in flax seed (secoisolariciresinol diglucoside or SDG). It is administered to research subjects in a product called BeneFlax, which a concentrated version of flax seed containing 38% SDG.

It is known that as people age, their bodies undergo physical changes both on the outside and the inside. The aging process may change the way that the investigators bodies deal with compounds the investigators eat. As an important measure of safety, the investigators want to check for evidence whether there is a difference in break down of SDG between different age groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults: 18-45 and 60-80 years of age

Exclusion Criteria:

* Strict vegetarians and vegans (as these diets likely contain foods which have higher levels of lignans)
* Strict vegetarians and vegans (as these diets likely contain foods which have higher levels of lignans)
* Individuals who smoke
* Individuals who have experienced diarrhea in the last three months
* Individuals who have taken oral antibiotics in the last three months
* Individuals who are currently taking warfarin or any of its derivatives
* Individuals with low haemoglobin (<121g/L for women and <137g/L for men)
* Individuals with BMI under 19 or over 28
* Pregnant or lactating women
* Women with child bearing potential not using contraceptives
* Current diagnosis of a bleeding disorder or at risk of bleeding
* Individuals with gastrointestinal problems (such as ulcers), or convulsive, depressive, or hepatic disorders
* Individuals with diabetes mellitus
* Individuals currently taking a flax seed supplement
* Individuals with an allergy to flax seed
* Individuals who have donated blood or lost > 450 mL of blood within 56 days of study duration
* Individuals who have participated in any other clinical trial with and investigational agent within one month of starting this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of secoisolariciresinol, enterodiol and enterolactone. | 0, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 72, 96 hours post-dose
  Blood samples will be collected at baseline and then post-dosing: every three hours for the first 48 hours, once at 72 hours and once at 96 hours. The concentrations of secoisolariciresinol, enterodiol and enterolactone will be quantitated at each time point.
Time to reach peak plasma concentration (tmax) of secoisolariciresinol, enterodiol and enterolactone. | 0, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 72, 96 hours post-dose
  Blood samples will be collected at baseline and then post-dosing: every three hours for the first 48 hours, once at 72 hours and once at 96 hours. The concentrations of secoisolariciresinol, enterodiol and enterolactone will be quantitated at each time point.
Area under the plasma concentration versus time curve (AUC) of secoisolariciresinol, enterodiol and enterolactone. | 0, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 72, 96 hours post-dose
  Blood samples will be collected at baseline and then post-dosing: every three hours for the first 48 hours, once at 72 hours and once at 96 hours. The concentrations of secoisolariciresinol, enterodiol and enterolactone will be quantitated at each time point.
Elimination rate constant (k) of secoisolariciresinol, enterodiol and enterolactone. | 0, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 72, 96 hours post-dose
  Blood samples will be collected at baseline and then post-dosing: every three hours for the first 48 hours, once at 72 hours and once at 96 hours. The concentrations of secoisolariciresinol, enterodiol and enterolactone will be quantitated at each time point.
Terminal phase half-life of secoisolariciresinol, enterodiol and enterolactone. | 0, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 72, 96 hours post-dose
  Blood samples will be collected at baseline and then post-dosing: every three hours for the first 48 hours, once at 72 hours and once at 96 hours. The concentrations of secoisolariciresinol, enterodiol and enterolactone will be quantitated at each time point.

SECONDARY OUTCOMES:
Food frequency questionnaire | at 0 hours - prior to study commencement
  Background information about participants usual dietary choices will be collected once prior to study commencement.
Activity questionnaire | at 0 hours - prior to study commencement
  Background information about participants usual physical activities will be collected once prior to study commencement.
Inflammatory markers | at 0 hours - prior to study commencement
  Measurement of the inflammatory markers interleukin-1a, interleukin-1b, interleukin-6 and TNF-a to determine participants baseline levels. The levels will only be tested once prior to study commencement

CONTACTS AND LOCATIONS:
Overall Officials: Jane Alcorn, DVM, PhD, Principal Investigator — College of Pharmacy & Nutrition, University of Saskatchewan
Locations (1):
- Saskatoon Centre for Patient Oriented Research - Saskatoon City Hospital, Saskatoon, Saskatchewan, Canada